CLINICAL TRIAL: NCT01753076
Title: Study NOG112264, a Phase II Study of Ozanezumab (GSK1223249) Versus Placebo in the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Study of Ozanezumab (GSK1223249) Versus Placebo in the Treatment of Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 112264
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; efficacy; ozanezumab; safety
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ozanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ozanezumab IV (Experimental): Administered by IV route. Treatment period - 48 Weeks
  Interventions: Drug: Ozanezumab
- Placebo (Placebo Comparator): Normal saline by IV route. Treatment period - 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozanezumab — Ozanezumab injection solution
  Arms: Ozanezumab IV
Drug: Placebo — Normal saline (0.9% sodium chloride) infusion
  Arms: Placebo

SUMMARY:
This is a 48-week, randomised, multi-centre, double-blind, placebo-controlled, parallel group investigation of the efficacy and safety of intravenous (IV) ozanezumab (GSK1223249) compared to placebo in subjects with Amyotrophic Lateral Sclerosis (ALS). Following a screening period of up to four weeks, eligible subjects will be randomised (1:1) to receive IV placebo or 15 milligram (mg)/ kilogram (kg) IV ozanezumab every 2 weeks for a period of 48 weeks with a follow-up visit around 14 weeks after the last infusion. A total of approximately 294 eligible subjects will be randomised from approximately 37 centers worldwide. The primary objective is to assess the effect of ozanezumab on the physical function and survival of ALS subjects over a treatment period of 48 weeks. Function will be measured using the ALS Functional Rating Scale - Revised (ALSFRS-R). Secondary objectives include the evaluation of other clinical outcomes associated with ALS (respiratory function, muscle strength, progression free survival and overall survival) in support of the primary objective. Quality of life, safety, tolerability, immunogenicity and pharmacokinetics (ozanezumab and riluzole) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of familial or sporadic ALS
* Onset of muscle weakness no more than 30 months before screening visit.
* Slow Vital Capacity (SVC) of at least 65% predicted for gender, age, ethnicity and height at Screening.
* If on riluzole, the dose must have been stable for at least 28 days prior to Baseline visit.
* Age 18 - 80 years inclusive.
* Female subjects may participate if they are of non-child-bearing potential or if they are of child-bearing potential they must agree to use the approved contraceptive methods
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2x upper limit of normal (ULN); alkaline phosphatase and bilirubin <=1.5xULN.
* QTc (both QTcB and QTcF) <450 milliseconds (msec) or <480 msec for subjects with Bundle Branch Block at Screening and Baseline (average from triplicate ECGs).

Exclusion Criteria:

* Patients with other neuromuscular disorders (including a history of polio) which in the opinion of the investigator could have contributed to the muscular atrophy or weakness caused by ALS
* Patients with primary lateral sclerosis, monomelic ALS, ALS Parkinsonism dementia complex.
* Patients requiring non-invasive or mechanical ventilation (non-invasive ventilation for sleep apnoea is allowed subject to discussion with Medical Monitor)
* Patients on diaphragmatic pacing.
* Presence of any of the following clinical conditions: Drug abuse or alcoholism, uncontrolled hypertension, active major infectious disease, unstable psychiatric illness within 90 days of the Screening visit
* Subjects, who in the investigator's judgement, pose a significant suicide risk. - Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), positive Hepatitis B surface antigen or Hepatitis C antibody test.
* Subjects who have participated in a clinical trial involving receipt of a biopharmaceutical product within 6 months prior to the first dosing day.
* Exposure to non-biological experimental agents 1 month or 5 half-lives prior to Baseline visit (whichever is longer).
* History of sensitivity to ozanezumab, or components thereof, or a history of other allergies that, in the opinion of the investigator, contraindicates participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- United States (4):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Columbus, Ohio
- Australia (2):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Herston, Queensland
- GSK Investigational Site, Leuven, Belgium
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (5):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
- Germany (6):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
- Italy (2):
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Verona, Veneto
- Japan (3):
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
- GSK Investigational Site, Utrecht, Netherlands
- GSK Investigational Site, Seoul, South Korea
- United Kingdom (3):
  - GSK Investigational Site, Preston, Lancashire
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Edgbaston

REFERENCES:
- [Derived] Meininger V, Genge A, van den Berg LH, Robberecht W, Ludolph A, Chio A, Kim SH, Leigh PN, Kiernan MC, Shefner JM, Desnuelle C, Morrison KE, Petri S, Boswell D, Temple J, Mohindra R, Davies M, Bullman J, Rees P, Lavrov A; NOG112264 Study Group. Safety and efficacy of ozanezumab in patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Neurol. 2017 Mar;16(3):208-216. doi: 10.1016/S1474-4422(16)30399-4. Epub 2017 Jan 28. PMID 28139349

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 304 participants were randomized (151 to placebo; 153 to ozanezumab 15 milligrams [mg]/kilogram [kg]), and 303 participants (151 placebo; 152 ozanezumab 15 mg /kg ) received at least one dose of investigational product (one of the participants who did not receive any study drug was re-randomized to ozanezumab).
Groups:
- Placebo: Participants (par) received placebo once every 2 weeks by intravenous infusion up to Week 46.
- Ozanezumab 15 mg/kg: Participants received ozanezumab 15 milligrams per kilogram (mg/kg) once every 2 weeks by intravenous infusion up to Week 46.
Period: Overall Study
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Started | 151 | 152
Completed | 110 | 106
Not Completed | 41 | 46
Not completed — Adverse Event | 17 | 18
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 4 | 2
Not completed — Withdrawal by Subject | 14 | 24
Not completed — Other-Reached Protocol-defined Stopping | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant who did not receive any study drug was excluded from the intent-to-treat (ITT) population.
Groups:
- Placebo: Participants received placebo once every 2 weeks by intravenous infusion up to Week 46.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ozanezumab 15 mg/kg | Total
Number analyzed (Participants) | 151 | 152 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (11.04) | 55.7 (10.40) | 55.6 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 49 | 103
  Male | 97 | 103 | 200
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 2 | 3
  Asian - Central/South Asian Heritage | 2 | 3 | 5
  Asian - East Asian Heritage | 3 | 8 | 11
  Asian - Japanese Heritage | 5 | 10 | 15
  Asian - South East Asian Heritage | 13 | 5 | 18
  White - Arabic/North African Heritage | 3 | 2 | 5
  White - White/Caucasian/European Heritage | 124 | 121 | 245
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Joint Rank Scores for Combined Analysis of Function (Amyotrophic Lateral Sclerosis Functional Rating Scale Revised [ALSFRS-R] Score) and 48 Week Overall Survival
Description: The joint rank score is a combined assessment of function and survival. Function is assessed using change from Baseline in the ALSFRS-R total score. To calculate joint rank scores, every participant was compared with all other participants in a pair wise manner and assigned a score of -1, 0 or 1 based on their relative outcomes. A subject's joint rank score is the sum of their scores across the pair wise comparisons. The . The ALSFRS-R was a quickly administered (5 min) ordinal rating scale used to determine a participant's assessment of their capability and independence in 12 functional activities. There were 12 questions, graded by the participant 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing. Lower scores of ALSFRS-R reflect greater impairment.
Time Frame: Week 48
Population: ITT population. Only on-treatment data (data within 21 days of the last dose) were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Placebo: Participants received placebo once every 2 weeks by intravenous infusion up to Week 46. Final outcome assessment conducted at Week 48.
- Ozanezumab 15 mg/kg: Participants received ozanezumab 15 milligrams per kilogram (mg/kg) once every 2 weeks by intravenous infusion up to Week 46. Final outcome assessment conducted at Week 48.
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 151 | 152
Scores on a scale | 15.0 (13.58) | -14.9 (13.54)
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.120, ANCOVA; Mean Difference (Final Values) = -30.0, 95% CI 2-sided [-67.9 to 7.9] — A negative mean difference means that the direction of effect is in favor of placebo

2. Secondary Outcome: Change From Baseline in the ALSFRS-R Total Score at Week 48
Description: The rate of decline was estimated by the change from Baseline in ALSFRS-R. The monthly slope for the ALSFRS-R score (i.e., the monthly rate of decline) was calculated as change from Baseline in the ALSFRS-R score at the last visit for that treatment period divided by the study day at the last visit for that treatment period /30.4. The Week 0 (Visit 2) value was considered to be the Baseline value. Change from Baseline was calculated by subtracting the derived Baseline value from the post-Baseline value. The ALSFRS-R was a quickly administered (5 min) ordinal rating scale used to determine a participant's assessment of their capability and independence in 12 functional activities. There were 12 questions, graded by the participant 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
Time Frame: Baseline and Week 48
Population: ITT Population. Only on-treatment data (data within 21 days of the last dose) were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 104 | 101
Scores on a scale | -9.1 (0.64) | -10.4 (0.64)
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.139, Mixed Models Analysis; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.1 to 0.4]

3. Secondary Outcome: Rate of Decline Over Week 48 in the ALSFRS-R Total Score
Description: The rate of decline was estimated by the change from Baseline in ALSFRS-R. The monthly slope for the ALSFRS-R score (i.e., the monthly rate of decline) was calculated as change from Baseline in the ALSFRS-R score at the last visit for that treatment period divided by the study day at the last visit for that treatment period devided by 30.4. The Week 0 (Visit 2) value was considered to be the Baseline value. Change from Baseline was calculated by subtracting the derived Baseline value from the post-Baseline value. The ALSFRS-R was a quickly administered (5 min) ordinal rating scale used to determine a participant's assessment of their capability and independence in 12 functional activities. There were 12 questions, graded by the participant 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
Time Frame: Baseline to Week 48
Population: ITT Population. Only on-treatment data (data within 21 days of the last dose) were analyzed..
Measure: Least Squares Mean (Standard Error); unit: change in scores on a scale per month
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 149 | 150
change in scores on a scale per month | -0.84 (0.063) | -0.96 (0.062)
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.173, Random coefficients analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.30 to 0.05]

4. Secondary Outcome: Change From Baseline in Slow Vital Capacity (SVC) at Week 48
Description: SVC was measured by using a validated spirometer. Three SVC measurements were performed for each participant at each assessment provided the difference from the second trial (if arranged by the numerical value) was not greater than 10%. If the difference between the best and the next best (based on the largest numerical value) SVC value from the first three trials was greater than 10%, additional trials (up to 5 in total) could have been performed. The Week 0 (visit 2) value was considered to be the Baseline value. Change from Baseline was calculated by subtracting the derived Baseline value from the post-Baseline value. A mixed-model repeated measures (MMRM) adjusted for treatment, visit, treatment by visit, Baseline SVC, Baseline SVC by visit, riluzole use. and country group was used for the analysis.
Time Frame: Baseline and Week 48
Population: ITT population. Only those participants available at indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 96 | 98
Liters (L) | -0.899 (0.0804) | -1.026 (0.0804)
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.265, Mixed Models Analysis; Mean Difference (Final Values) = -0.127, 95% CI 2-sided [-0.351 to 0.097]

5. Secondary Outcome: Change From Baseline in Muscle Strength as Measured by Hand Held Dynamometry (HHD) Score at Week 48
Description: The HHD is a device placed between the hand of the practitioner and the tested body part and provides a quantified measurement of muscle strength. Each muscle was tested twice, and both values were recorded. Additionally, a third trial could have been performed if the variability between the first two trials was greater than 15 % or if the rater thought that one of the first two trials was not valid. The Week 0 (Visit 2) value was considered to be the Baseline value. Percent change from Baseline for each muscle group was calculated as 100*(HHD score minus the Baseline score) divided by the Baseline score. The average percent change was the mean percent change across the muscle groups that were non-missing/non-zero at Baseline. MMRM adjusted for treatment, visit, treatment by visit, number of non-missing/non-zero muscle groups at Baseline, number of non-missing/non-zero muscle groups at Baseline by Visit, riluzole use, and country group was used for the analysis.
Time Frame: Baseline and Week 48
Population: ITT Population. Only participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 99 | 95
Percent change | -34.7 (3.77) | -42.9 (3.75)
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.125, Mixed Models Analysis; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-18.7 to 2.3]

6. Secondary Outcome: Number of Clinical Global Impression-improvement Scale (CGI-I) Responders at Week 48
Description: The CGI-I scale is a single observer-rated item measuring global improvement relative to Baseline. The CGI-I score is rated on a 7-point scale, from 1 (very much improved) to 7 (very much worse). Participant status at Baseline was assessed using the Clinical Global Impression Severity scale (CGI-S), which is a 7-point scale (1: normal, not at all ill; 7: most extremely ill) used to rate the severity of the participant's illness. Participants achieving a score of 1-4 in the CGI-I at Week 48 were considered to be responders. A a logistic regression adjusted for CGI-S at Baseline, riluzole use, and world region was used for the analysis.
Time Frame: Week 48
Population: ITT Population. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 101 | 97
Participants | 23 | 18
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.393, Regression, Logistic; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.36 to 1.49]

7. Secondary Outcome: Overall Survival at Week 48 and Week 60
Description: Overall survival is defined as the time from randomization to death or censoring at the time point of analysis, whichever comes first. Kaplan Meier estimates at Week 48 were evaluated at Day 344. A participant was considered to have completed if he/she was censored at Day 344. Kaplan Meier estimates at Week 60 were evaluated at Day 428. A participant was considered to have completed if he/she was censored at Day 428. Confidence intervals were estimated using the Brookmeyer Crowley method. Results are shown as the estimated percentage of participants alive at Weeks 48 and 60. Week 48: Only on-treatment data (data within 21 days of the last dose) were analyzed. Week 60: Including off treatment data (data after 21 days after the last dose) were analyzed.
Time Frame: Week 48 and Week 60
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo: Participants received placebo once every 2 weeks by intravenous infusion up to Week 46. Outcome assessments conducted at Week 48 and Week 60.
- Ozanezumab 15 mg/kg: Participants received ozanezumab 15 mg/kg once every 2 weeks by intravenous infusion up to Week 46. Outcome assessments conducted at Week 48 and Week 60.
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 151 | 152
Percentage of participants
  Week 48 | 95.5 [92.0 to 99.0] | 94.3 [90.4 to 98.1]
  Week 60 | 87.4 [81.5 to 93.3] | 85.4 [79.4 to 91.3]
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.986, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.34 to 2.89] — Week 48
Statistical Analysis 2: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.923, Chi-squared; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.53 to 2.01] — Week 60

8. Secondary Outcome: Progression-free Survival at Week 48
Description: Progression-free survival at Week 48 is defined as the time from randomization to progression (decline of at least six points on the ALSFRS-R from Baseline) or death or censored at Week 48, whichever comes first. Kaplan Meier estimates at Week 48 were evaluated at Day 344. A participant was considered to have completed if he/she was censored at Day 344. Confidence intervals were estimated using the Brookmeyer Crowley method. Results are shown as the estimated percentage of participants alive and without disease progression at Week 48.
Time Frame: Week 48
Population: ITT Population. Only on-treatment data (data within 21 days of the last dose) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants surviving
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 151 | 152
Percentage of participants surviving | 30.8 [23.0 to 38.6] | 28.5 [21.1 to 35.9]
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; p = 0.642, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.81 to 1.42]

9. Secondary Outcome: Change From Baseline in the EuroQol 5 Dimensions-5 Level Short Form (EQ-5D-5L) Utility Score at Week 48
Description: A utility score for each participant was calculated based on the value set for England. The Week 0 (Visit 2) value was considered to be the Baseline value. Change from Baseline was calculated by subtracting the derived Baseline value from the post-Baseline value. EQ-5D-5L is a standardized, participant-rated instrument for use as a measure of health outcomes. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the EQ-Visual Analog Scale (EQ-VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). . For each of these dimensions, the participant self assigned a score: 1 (no problems); 2 (slight problems); 3 (moderate problems); 4 (severe problems); 5 (extreme problems).Minimum score on scale was 1 and maximum score was 5 for each dimension. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 48
Population: ITT Population. Only participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 103 | 102
Scores on a scale | -0.234 (0.0207) | -0.238 (0.0207)
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.062 to 0.053]

10. Secondary Outcome: Change From Baseline in the Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) Total Score at Week 48
Description: The ALSAQ-40 is a disease specific health status assessment for individuals with ALS/motor neuron disease. The ALSAQ-40 is comprised of 40 questions measuring 5discrete dimensions of health status that are affected by the disease: physical mobility (10 items); activities of daily living and independence (10 items); eating and drinking (3 items); communication (7 items); emotional reactions (10 items). Participants were asked to indicate the frequency of each event by selecting one of five options (Likert scale: 0-4): never/rarely/sometimes/often/ always or cannot do at all. The total score (minimum possible score=0, maximum possible score=160) was calculated by adding the five domain scores. A low score indicates a better health state. Change from Baseline was calculated by subtracting the derived Baseline value from the post-Baseline value. A mixed-model repeated measures adjusted for treatment, Visit, Treatment by Visit, and Baseline ALSAQ-40 total score was used for the analysis.
Time Frame: Baseline and Week 48
Population: ITT Population. Only participants with data available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Ozanezumab 15 mg/kg
Number analyzed (Participants) | 102 | 96
Scores on a scale | 19.2 (1.47) | 20.6 (1.49)
Statistical Analysis 1: Comparison: Placebo vs Ozanezumab 15 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-2.8 to 5.5]

ADVERSE EVENTS:
Time Frame: Up to Week 64
Description: AEs and SAEs were collected in members of the Safety Population, comprised of all participants in the treatment cohort who gave informed consent, were randomized, and received at least one dose of study medication.
Groups:
- Ozanezumab IV: Participants received ozanezumab 15 mg/kg once every 2 weeks by intravenous infusion up to Week 46.
Arm/Group | Placebo | Ozanezumab IV
All-Cause Mortality (participants affected / at risk) | 13/151 | 18/152
Serious Adverse Events (participants affected / at risk) | 46/151 | 47/152
Other Adverse Events (participants affected / at risk) | 119/151 | 120/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Ozanezumab IV (N=152)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Eye penetration (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Motor neurone disease (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Parosmia (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2
Catheter site pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Euthanasia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 2 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Ozanezumab IV (N=152)
Fall (Injury, poisoning and procedural complications) | 68 | 56
Contusion (Injury, poisoning and procedural complications) | 18 | 11
Diarrhoea (Gastrointestinal disorders) | 12 | 25
Constipation (Gastrointestinal disorders) | 12 | 23
Nausea (Gastrointestinal disorders) | 11 | 14
Dyspepsia (Gastrointestinal disorders) | 4 | 10
Vomiting (Gastrointestinal disorders) | 8 | 5
Nasopharyngitis (Infections and infestations) | 32 | 35
Urinary tract infection (Infections and infestations) | 10 | 5
Bronchitis (Infections and infestations) | 8 | 6
Headache (Nervous system disorders) | 26 | 29
Dizziness (Nervous system disorders) | 14 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 11
Fatigue (General disorders) | 13 | 11
Oedema peripheral (General disorders) | 12 | 12
Peripheral swelling (General disorders) | 7 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 17
Anxiety (Psychiatric disorders) | 9 | 7
Depression (Psychiatric disorders) | 5 | 11
Haematoma (Vascular disorders) | 10 | 5
Hypertension (Vascular disorders) | 8 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.